CLINICAL TRIAL: NCT04519957
Title: Multicentre Study To Assess Safety And Efficacy Of Psilocybin In Patients With Treatment-Resistant Depression Following Completion Of COMP 001 And COMP 003 Trials (P-TRD LTFU)
Brief Title: Long Term Follow Up Study to COMP 001 And COMP 003 Trials (P-TRD LTFU)
Status: Completed | Type: Observational
Sponsor: COMPASS Pathways (Industry)
Responsible Party: Sponsor
Other Study IDs: COMP004
Record Dates: First submitted 2020-08-13; First posted 2020-08-20 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to assess the long-term efficacy of psilocybin with respect to use of new antidepressant treatment, hospitalisations for depression, suicidality, and depressive severity rated using the Montgomery and Asberg Depression Rating Scale (MADRS) over a total of 52 weeks (compared across the 1 mg, 10 mg and 25 mg psilocybin groups from COMP 001).

DETAILED DESCRIPTION:
In this present study (COMP 004), the aim is to follow up participants from COMP 001 and COMP 003 in a long-term follow up study, with both remote and digital assessments, to explore the long term efficacy and safety of the three different doses of psilocybin (1 mg, 10 mg, and 25 mg) administered to patients with TRD as a monotherapy in COMP 001 and 25 mg psilocybin administered as an adjunct to an SSRI in COMP 003. Patients previously treated in COMP001 will be followed for approximately 40 weeks and patients previosuly treated in COMP003 will be followed for approximately 49 weeks giving a total follow up period of 52 weeks from psilocybin dosing.

ELIGIBILITY:
Inclusion Criteria:

Signed ICF Each participant having completed the final study visit of either COMP 001 or COMP 003 Ability to complete all protocol required assessment tools (including having access to the internet in order to complete the digital assessments) without any assistance or alteration to the copyrighted assessments, and to comply with all study visits

Exclusion Criteria:

Subject has any condition, for which in the opinion of the investigator, participation would not be in the interest of the subject eg participation could compromise the wellbeing of the participant or prevent, limit, or confound the protocol-specified assessments

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: TRD patients who completed COMP001 or COMP003
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Long-term efficacy of psilocybin | up to 52 weeks
  Use of new antidepressant treatment, hospitalisations for depression, suicidality, and depressive severity rated using the Montgomery and Asberg Depression Rating Scale (MADRS)

SECONDARY OUTCOMES:
Response, sustained response, remission and change in depression severity | Up to 52 weeks
  Montgomery Asberg Depression Rating Scale (MADRS)
Psychosocial functioning and to predict durability of response to antidepressant treatment | up to 52 weeks
  Work and Social Adjustment Scale (WSAS) score change from Baseline of the prior study
Functional impairment in work/school, social life, and family life. | Up to 52 weeks
  Sheehan Disability Scale (SDS) score change from Baseline of the prior study
Safety of Psilocybin | Up to 52 weeks
  Incidence and severity of Adverse Events (AEs) and Seroius Adverse Events (SAEs)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (4):
  - Kadima Neuropsychiatry Institute, La Jolla, California
  - Altman Clinical and Translational Research Institute, University of California, San Diego, California
  - Mood and Anxiety Disorders Program Emory University School of Medicine, Atlanta, Georgia
  - UT Center of Excellence on Mood Disorders, University of Texas Health Science Center, Houston, Texas
- National Institute of Mental Health Czech Republic, Klecany, Czechia
- Sheaf House, Tallaght Hospital, Dublin, Ireland
- Groningen University Medical Centre, Groningen, Netherlands
- Kings College London, Institute of Psychiatry, Psychology and Neurology, London, United Kingdom

REFERENCES:
- [Derived] Goodwin GM, Nowakowska A, Atli M, Dunlop BW, Feifel D, Hellerstein DJ, Marwood L, Shabir Z, Mistry S, Stansfield SC, Teoh E, Tsai J, Young MB, Malievskaia E. Results From a Long-Term Observational Follow-Up Study of a Single Dose of Psilocybin for a Treatment-Resistant Episode of Major Depressive Disorder. J Clin Psychiatry. 2025 Mar 3;86(1):24m15449. doi: 10.4088/JCP.24m15449. PMID 40047545